CLINICAL TRIAL: NCT07141563
Title: Retrospective Study for Describing Real-World Effectiveness of Nivolumab + Chemotherapy in Neoadjuvant NSCLC in Argentina
Brief Title: A Study Describing Real-World Effectiveness of Nivolumab + Chemotherapy in Neoadjuvant NSCLC
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Grupo Argentino Oncología Torácica (GAOT) - Asociación Argentina Oncología Clínica (AAOC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CA209-1524
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Platinum Compounds; Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; Gemcitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with resectable non-small cell lung cancer (NSCLC) receiving neoadjuvant treatment with nivolumab in combination with platinum-based chemotherapy
  Interventions: Drug: Nivolumab + platinum-based chemotherapy

INTERVENTIONS:
Drug: Nivolumab + platinum-based chemotherapy — According to the product label
  Other Names: Opdivo, Cisplatin, Carboplatin, Pemetrexed, Paclitaxel, Gemcitabine.

SUMMARY:
The purpose of this study is to evaluate the real-world effectiveness and safety of neoadjuvant nivolumab combined with chemotherapy in Argentinian patients with resectable non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This is a non-interventional, retrospective, single-arm, multicenter study evaluating the real-world effectiveness of neoadjuvant nivolumab plus platinum-based chemotherapy in Argentinian patients with resectable non-small cell lung cancer (NSCLC). The primary objective is to estimate the rate of pathological complete response (pCR) following neoadjuvant therapy.

Adult patients (≥18 years) with newly diagnosed, early-stage, resectable NSCLC (stage IIA-IIIB, AJCC 8th ed) and no EGFR or ALK driver mutations who initiated neoadjuvant nivolumab (360 mg Q3W) plus platinum-based chemotherapy between July 1, 2022, and March 1, 2025, at participating Argentinian centers will be included. Data will be extracted retrospectively from medical records for up to 12 months following surgery or neoadjuvant therapy.

The primary endpoint is the pathological complete response (pCR), defined as absence of residual viable tumor in both lung and lymph nodes at surgery. Secondary endpoints include major pathological response (MPR), event-free survival (EFS) over 1 year, surgical outcomes, safety, and subsequent adjuvant therapy use. Descriptive and survival analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older
* Participants diagnosed with resectable non-small cell lung cancer (NSCLC) (stage IIA-IIIB TNM AJCC 8ed) according to the treating team's judgment
* Participants who received nivolumab and chemotherapy as neoadjuvant therapy between 1st July 2022 and 1st March 2025
* Participants must have given informed consent for their data to be used for research or academic studies, or a waiver of consent has been obtained

Exclusion Criteria:

* Participants with confirmed positive EGFR gene mutation or ALK fusion gene, as the study focuses on the effectiveness of nivolumab in patients without these driver mutations
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Participants who received any antineoplastic therapy within 3 months prior to initiating neoadjuvant nivolumab and chemotherapy, to avoid confounding effects from prior treatments
* Participants who participated in a clinical trial for NSCLC, to ensure the study reflects real-world clinical practice
* Participants with complications of treatment-related adverse events related to hematotoxicity of antineoplastic agents 3 months prior to the start of neoadjuvant therapy, to minimize risks and confounding factors
* Participants who started neoadjuvant therapy outside the participating medical institution and were transferred to the institution for surgery, to ensure data consistency and reliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults diagnosed with resectable non-small cell lung cancer (NSCLC) and have undergone neoadjuvant treatment with nivolumab in combination with platinum-based chemotherapy according to routine clinical practice in Argentina between 1st July 2022 and 1st March 2025
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Rate of pathological complete response (pCR) post-surgery | Up to 1 year
  Number of patients with complete pathological response (defined as absence of residual viable tumor in both lung and lymph nodes at surgery) divided by total number of patients.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 1 year
  Defined as the time from the start of neoadjuvant therapy to the occurrence of any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause
Rate of major pathological response (MPR) post-surgery | Up to 1 year
  Proportion of patients with less than 10% residual viable tumor after neoadjuvant therapy, assessed at surgery.
Participant demographics | Baseline
  Socio-demographic characteristics of patients, such as age, sex and tobacco use.
Participant clinical characteristics | Baseline
  Clinical characteristics of patients, describing the proportion and characteristics of patients who receive adjuvant RT and/or CT as subsequent treatment, and assessing surgical outcomes and adverse events (AEs)
Number of participants receiving surgery | Up to 1 year
  Number of patients receiving surgery after neoadjuvant treatment
Time from diagnosis to neoadjuvant treatment start before surgery | Up to 1 year
  Discrete dates difference
Number of nivolumab doses received before surgery | Up to 1 year
  Continues variable
Type of chemotherapy given in combination to nivolumab adjuvant treatment before surgery | Up to 1 year
  Drugs received: Cisplatin, Carboplatin Pemetrexed, Paclitaxel, Gemcitabine
Relapse status | Up to 1 year
  Date of investigator-assessed relapse and type of relapse (Locoregional, Distant)
Surgery type | Up to 1 year
  Surgical approach (thoracotomy, VATS or robotic thoracic surgery) and surgical procedure type (lobectomy, segmentectomy, wedge resection, or pneumonectomy) will be recorded at the time of surgery.
Extent of surgical resection | Up to 1 year
  R0, R1, R2
Surgical complications during or after surgery | Up to 1 year
  Pre-established categories or categories formed based on free-text information available.
Reasons for not having surgery | Up to 1 year
  ECOG Performance Status > 1, Major associated pathologies that increase the surgery risk to an unacceptable level, Disease progression, Adverse event Toxicity, Patient refusal, Poor lung function, Unresectability, Death, Others
Treatment received after neoadjuvant treatment | Up to 1 year
  Treatment subsequent to neoadjuvant therapy, including radiotherapy, chemotherapy, immuno-oncology therapy, targeted therapy, or other treatments, will be recorded with treatment start and end dates during follow-up.
Reason for having adjuvant treatment | Up to 1 year
  Pre-established categories or categories formed based on free-text information available
Adverse events (AEs) | Up to 1 year
  Describe the frequency and severity of AEs and IMAEs, including intensity, seriousness, causality, preferred terms, organ class and event outcome.
  Analyses will be performed at both patient-level and at event-level overall, by intensity and by causality. For the patient-level analysis, patients will be counted once by AE considering the maximum grade.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Perfetti, MD, Principal Investigator — Asociación Argentina Oncología Torácica (AAOC); Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Grupo Argentino Oncología Torácica (GAOT) - Asociación Argentina Oncología Clínica (AAOC), Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts